CLINICAL TRIAL: NCT00780624
Title: Nasal Intermittent Positive Pressure Ventilation In Newborn Infants With Respiratory Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yuan Shi, Professor and Chief of Pediatrics, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCR2008053
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Respiratory Distress Syndrome
Keywords: RDS; Infant, newborn; NIPPV; CPAP
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIPPV (Active Comparator): The NIPPV group receiving NIPPV treatment.
  Interventions: Device: NIPPV
- Control (Active Comparator): The Control group receiving nCPAP treatment.
  Interventions: Device: NIPPV

INTERVENTIONS:
Device: NIPPV — Ventilator is Bird VIP.
Device: NIPPV — Ventilator(Bird VIP) is used for NIPPV device. Non-invasive NIPPV is used in the NIPPV group instead of nCPAP in the control group.
Device: NIPPV — Ventilator (Bird VIP, USA) is used for provide of NIPPV in the NIPPV group instead of nCPAP in the control group. The duration of NIPPV is according to the baby's respiratory condition.

SUMMARY:
The submitted trial is the first prospective, randomized trial comparing nasal intermittent positive pressure ventilation(NIPPV) vs nCPAP in newborn infants with respiratory distress syndrome.

DETAILED DESCRIPTION:
Nasal intermittent positive pressure ventilation (NIPPV) is similar to nCPAP, but also gives some breaths, or extra support, to newborn infants through a small tube in the nose. NIPPV is safe and effective, and already in use as an alternate "standard" therapy. Nevertheless, NIPPV has never been used in chinese babies.

The submitted trial is the first prospective, randomized trial Comparing NIPPV vs nCPAP in newborn infants with respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Newborn infants with birth weight >500 gm.
2. Gestational age >24 completed weeks.
3. Intention to manage the infant with non-invasive respiratory support (i.e. no endotracheal tube), where either: 1) the infant is within the first 7 days of life and has never been intubated or has received less than 24 hours of total cumulative intubated respiratory support; 2)the infant is within the first 28 days of life, has been managed with intubated respiratory support for 24 hours or more and is a candidate for extubation followed by non-invasive respiratory support.
4. No known lethal congenital anomaly or genetic syndromes.
5. Signed parental informed consent.

Exclusion Criteria:

1. Considered non-viable by clinician (decision not to administer effective therapies)
2. Life-threatening congenital abnormalities including congenital heart disease (excluding patent ductus arteriosis)
3. Infants known to require surgical treatment
4. Abnormalities of the upper and lower airways
5. Neuromuscular disorders
6. Infants who are >28 days old and continue to require mechanical ventilation with an endotracheal tube

Ages: 1 Minute to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Mechanical Ventilation via endotracheal tube after non-invasive respiratory support. | At 7 days after non-invasive respiratorynsupport.

SECONDARY OUTCOMES:
Overall clinical outcomes at 7 days, 28 days, and 36 weeks postmenstrual age. | At 7 days, 28 days and at 36 weeks postmenstraul age

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shi, MD, Study Director — Department of Pediatrics, Daping Hospital, Third Military Medical University
Locations (1):
- Deaprtment of Pediatrics, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shi Y, Tang S, Zhao J, Shen J. A prospective, randomized, controlled study of NIPPV versus nCPAP in preterm and term infants with respiratory distress syndrome. Pediatr Pulmonol. 2014 Jul;49(7):673-8. doi: 10.1002/ppul.22883. Epub 2013 Sep 4. PMID 24039148